CLINICAL TRIAL: NCT06534034
Title: Clinical Outcome of Dentsply Sirona Profile Implants: A 12-year Follow-up Retrospective Study.
Brief Title: Clinical Outcome of Dentsply Sirona Profile Implants
Status: Completed | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: RETROPROF
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Dental Implants
Keywords: Dental Implant; Complication; Astra Tech Osseospeed Profile
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Astra Tech Profile: Patients who has receive Astra Tech Profile dental implant system placement.
  Interventions: Procedure: Dental implant placement

INTERVENTIONS:
Procedure: Dental implant placement — Dental implant placement on edentulous jaw.
  Other Names: implant surgery; implant prosthesis

SUMMARY:
This is a retrospective observational study of 50 implants placed between 2013 and 2023 from the same dental implant system (Osseospeed Profile, Dentsply Implants, Mölndal, Sweden).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the cumulative survival, success and complication rates obtained with the use of Osseospeed Profile EV implants in two clinical centres with similar characteristics since its launch on the market in 2013, until today.

All clinical records of patients with this implant system will be collected and the following data will be recorded:

Patient gender Date of placement Dimensions and location of implant(s) placed Type of implantation Design of the implant-supported dental prosthesis, single or partial, screw-retained or cemented Date of last radiographic control Type of biological and/or mechanical complications that occurred In biological complications, presence or absence of inflammatory signs and presence or absence of peri-implant bone loss.

For mechanical complications, screw loosening, porcelain fracture, fracture of the prosthetic abutment or fracture of the implant.

Date of explantation if present

The mean, standard deviation (SD), and percentage will be calculated for all recorded parameters.

A life table will be made with cumulative survival and success rate (CSR), according to Kaplan-Meier analysis. Correlations and regression analysis will be performed to assess the influence of the variables on the outcomes

Conclusions will be drawn based on the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have come to private dental clinics with the need to rehabilitate a single edentulous space in the posterior mandibular area.

Exclusion Criteria:

* None

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who receive Astra Tech Osseospeed Profile dental implant system placement at two private dental clinics in Spain.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Success Rate | through study completion, a maximum of 5 years
  Number of dental Implants in function with no complications events
Survival Rate | through study completion, a maximum of 5 years
  Number of dental Implants in function with any complications events

SECONDARY OUTCOMES:
Biological complications rate | through study completion, a maximum of 5 years
  Number os dental implant treatment with some biological complication
Mechanical complications rate | through study completion, a maximum of 5 year
  Number of dental implant treatment with some mechanical complication

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, PhD, Principal Investigator — Aula Dental Avanzada
Locations (2):
- Spain (2):
  - Clínica Dental Esteve, Alicante
  - Clinica Dental Amigó, Valencia

IPD SHARING:
Plan to Share IPD: No